CLINICAL TRIAL: NCT06683677
Title: High Flow Nasal Cannula is Appropriate Alternative for Stabilization of Extremely Premature Infants: a Prospective Observational Study
Brief Title: High Flow Nasal Cannula for Stabilization of Extremely Premature Infants
Acronym: SIMPLSAFE2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jonáš Klára, Principal Investigator, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16/24
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Premature Infant; Ventilation Therapy; High Flow Nasal Canula
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-flow-nasal-cannula (Experimental): Extremely preterm infants receive High-Flow Nasal Cannula therapy immediately after birth. The intervention includes placental transfusion, followed by administering High-Flow Nasal Cannula at a flow rate of 8 l/min along with intermittent tactile stimulation. Criteria for switching to Continuous Positive Airway Pressure or Positive Pressure Ventilation are established for cases of persistent bradycardia or low Saturation of oxygen (SpO2).
  Interventions: Device: High-Flow Nasal Cannula

INTERVENTIONS:
Device: High-Flow Nasal Cannula — The intervention involves administering High-Flow Nasal Cannula therapy to extremely preterm infants immediately after birth.

SUMMARY:
A prospective observational study evaluates the safety and efficacy of using High-Flow Nasal Cannula to stabilize extremely preterm infants immediately after birth. Following placental transfusion, high flow nasal cannula at 6-8 l/min is administered along with intermittent tactile stimulation. Criteria for switching to other interventions like continuous positive airway pressure or positive pressure ventilation are set for cases of persistent bradycardia or low Saturation of oxygen (SpO2).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 25+0 and 27+6 gestational weeks
* Weight above 500 grams

Exclusion Criteria:

* Previable rupture of membranes,
* Congenital malformations previable
* Acute intrauterine hypoxia.

Ages: 0 Minutes to 2 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Positive pressure ventilation after delivery | 10 minutes
  The number of infants who required positive pressure ventilation (PPV) in the first ten minutes after delivery.

SECONDARY OUTCOMES:
SpO₂ > 80% in five minutes after delivery | 5 minutes
  The number of infants with SpO₂ > 80% five minutes after delivery, with or without the use of positive pressure ventilation (PPV).
SpO₂ > 90% ten minutes after delivery | 10 minutes
  The number of infants with SpO₂ > 90% ten minutes after delivery without the use of positive pressure ventilation (PPV).

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital Prague, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manley BJ, Arnolda GRB, Wright IMR, Owen LS, Foster JP, Huang L, Roberts CT, Clark TL, Fan WQ, Fang AYW, Marshall IR, Pszczola RJ, Davis PG, Buckmaster AG; HUNTER Trial Investigators. Nasal High-Flow Therapy for Newborn Infants in Special Care Nurseries. N Engl J Med. 2019 May 23;380(21):2031-2040. doi: 10.1056/NEJMoa1812077. PMID 31116919
- [Background] Roberts CT, Owen LS, Manley BJ, Froisland DH, Donath SM, Dalziel KM, Pritchard MA, Cartwright DW, Collins CL, Malhotra A, Davis PG; HIPSTER Trial Investigators. Nasal High-Flow Therapy for Primary Respiratory Support in Preterm Infants. N Engl J Med. 2016 Sep 22;375(12):1142-51. doi: 10.1056/NEJMoa1603694. PMID 27653564
- [Background] Bjorland PA, Oymar K, Ersdal HL, Rettedal SI. Incidence of newborn resuscitative interventions at birth and short-term outcomes: a regional population-based study. BMJ Paediatr Open. 2019 Dec 29;3(1):e000592. doi: 10.1136/bmjpo-2019-000592. eCollection 2019. PMID 31909225
- [Background] Norman E, Westrin P, Fellman V. Placental transfer and pharmacokinetics of thiopentone in newborn infants. Arch Dis Child Fetal Neonatal Ed. 2010 Jul;95(4):F277-82. doi: 10.1136/adc.2009.177626. Epub 2010 May 20. PMID 20488867
- [Background] Tana M, Tirone C, Aurilia C, Lio A, Paladini A, Fattore S, Esposito A, De Tomaso D, Vento G. Respiratory Management of the Preterm Infant: Supporting Evidence-Based Practice at the Bedside. Children (Basel). 2023 Mar 10;10(3):535. doi: 10.3390/children10030535. PMID 36980093
- [Background] Diggikar S, Ramaswamy VV, Koo J, Prasath A, Schmolzer GM. Positive Pressure Ventilation in Preterm Infants in the Delivery Room: A Review of Current Practices, Challenges, and Emerging Technologies. Neonatology. 2024;121(3):288-297. doi: 10.1159/000537800. Epub 2024 Mar 11. PMID 38467119
- [Background] Foglia EE, Shah BA, Szyld E. Positive pressure ventilation at birth. Semin Perinatol. 2022 Oct;46(6):151623. doi: 10.1016/j.semperi.2022.151623. Epub 2022 May 21. PMID 35697527
- [Background] Roehr CC, Yoder BA, Davis PG, Ives K. Evidence Support and Guidelines for Using Heated, Humidified, High-Flow Nasal Cannulae in Neonatology: Oxford Nasal High-Flow Therapy Meeting, 2015. Clin Perinatol. 2016 Dec;43(4):693-705. doi: 10.1016/j.clp.2016.07.006. PMID 27837753
- [Background] Mazmanyan P, Darakchyan M, Pinkham MI, Tatkov S. Mechanisms of nasal high flow therapy in newborns. J Appl Physiol (1985). 2020 Apr 1;128(4):822-829. doi: 10.1152/japplphysiol.00871.2019. Epub 2020 Feb 20. PMID 32078463
- [Background] Roberts CT, Hodgson KA. Nasal high flow treatment in preterm infants. Matern Health Neonatol Perinatol. 2017 Sep 6;3:15. doi: 10.1186/s40748-017-0056-y. eCollection 2017. PMID 28904810
- [Background] Siva NV, Reynolds PR. Stabilisation of the preterm infant in the delivery room using nasal high flow: A 5-year retrospective analysis. Acta Paediatr. 2021 Jul;110(7):2065-2071. doi: 10.1111/apa.15824. Epub 2021 Mar 8. PMID 33638878
- [Background] Reynolds P, Leontiadi S, Lawson T, Otunla T, Ejiwumi O, Holland N. Stabilisation of premature infants in the delivery room with nasal high flow. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F284-7. doi: 10.1136/archdischild-2015-309442. Epub 2016 Jan 5. PMID 26733541
- [Background] Kuypers KLAM, Hopman A, Cramer SJE, Dekker J, Visser R, Hooper SB, Te Pas AB. Effect of initial and subsequent mask applications on breathing and heart rate in preterm infants at birth. Arch Dis Child Fetal Neonatal Ed. 2023 Nov;108(6):594-598. doi: 10.1136/archdischild-2022-324835. Epub 2023 Apr 20. PMID 37080734
- [Background] Kuypers K, Martherus T, Lamberska T, Dekker J, Hooper SB, Te Pas AB. Reflexes that impact spontaneous breathing of preterm infants at birth: a narrative review. Arch Dis Child Fetal Neonatal Ed. 2020 Nov;105(6):675-679. doi: 10.1136/archdischild-2020-318915. Epub 2020 Apr 29. PMID 32350064
- [Background] Martherus T, Oberthuer A, Dekker J, Hooper SB, McGillick EV, Kribs A, Te Pas AB. Supporting breathing of preterm infants at birth: a narrative review. Arch Dis Child Fetal Neonatal Ed. 2019 Jan;104(1):F102-F107. doi: 10.1136/archdischild-2018-314898. Epub 2018 Jul 26. PMID 30049727
- [Background] Lista G, Cavigioli F, La Verde PA, Castoldi F, Bresesti I, Morley CJ. Effects of Breathing and Apnoea during Sustained Inflations in Resuscitation of Preterm Infants. Neonatology. 2017;111(4):360-366. doi: 10.1159/000454799. Epub 2017 Jan 25. PMID 28118641
- [Background] Kirpalani H, Ratcliffe SJ, Keszler M, Davis PG, Foglia EE, Te Pas A, Fernando M, Chaudhary A, Localio R, van Kaam AH, Onland W, Owen LS, Schmolzer GM, Katheria A, Hummler H, Lista G, Abbasi S, Klotz D, Simma B, Nadkarni V, Poulain FR, Donn SM, Kim HS, Park WS, Cadet C, Kong JY, Smith A, Guillen U, Liley HG, Hopper AO, Tamura M; SAIL Site Investigators. Effect of Sustained Inflations vs Intermittent Positive Pressure Ventilation on Bronchopulmonary Dysplasia or Death Among Extremely Preterm Infants: The SAIL Randomized Clinical Trial. JAMA. 2019 Mar 26;321(12):1165-1175. doi: 10.1001/jama.2019.1660. PMID 30912836
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829